CLINICAL TRIAL: NCT05778383
Title: Zinc-based Nutritional Immunity to Lower Inflammation, Viral Load and COVID-19 Mortality During SARS-CoV-2 Infection.
Brief Title: Zinc Supplementation Impact in Acute COVID-19 Clinical Outcomes
Acronym: MARZINC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Universitat Pompeu Fabra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/9673/I
Record Dates: First submitted 2023-03-04; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2021-03

CONDITIONS: Zinc Deficiency; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Zinc Acetate

STUDY DESIGN:
Intervention Model Description: We are administering Zinc supplementation in the acute phase of SARS-CoV-2 infection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standars of Care (No Intervention): Standard of Care of treatment for SARS-coV-2 infection
- Zinc Supplementation +Standard of Care (Experimental): Standard of care + ( 240mg zinc acetate Zinc (75mg Zn element) +NM QD) during 14 days
  Interventions: Dietary Supplement: Zinc Acetate

INTERVENTIONS:
Dietary Supplement: Zinc Acetate — Each participant allocated in the intervention arm will be treated as Standard of Care and will be supplemented with 240mg of Zinc Acetate
  Arms: Zinc Supplementation +Standard of Care

SUMMARY:
Infections with SARS-CoV-2 result in a systemic disease with a variety of outcomes, from no symptoms to severe and diverse pathologies. Therefore, it is important to identify risk factors determining COVID-19 severity, especially if those factors might be adjusted, allowing early and effective therapeutic interventions. Zinc is a trace element essential for human health. Zinc deficiency is common in old adults, vegetarians and patients with chronic inflammatory diseases. This condition causes immune dysfunction leading to increased risk of inflammatory and infectious diseases, including acquired immune deficiency syndrome, measles, malaria, tuberculosis, and pneumonia. Besides, zinc has a direct antiviral activity against specific viruses like rhinovirus, HCV, herpes simplex virus. In this scenario, it has been shown that zinc supplementation has benefits on the recurrence and persistence of acute and chronic viral infections like common cold or HCV, HBV. Moreover, our team has recently done an observational study with 249 COVID-19 patients that showed how COVID-19 patients with lower plasma zinc content had worse prognosis, increased time of hospitalization and mortality.

Therefore, the main aim of the project is to explore the therapeutic benefit of zinc supplementation for COVID-19 patients and to determine the cellular and molecular basis of the effect of Zn levels on SARS CoV-2 infections. For that purpose the investigators will run a clinical trial supplementing with zinc COVID-19 patients. Moreover, the investigators will carry out experiments to understand the association between zinc nutritional status and SARS-Cov-2 infection progression in cellular and animal models.

Given the current knowledge about zinc supplementation toxicity and dosage, the investigators expect that recommendations derived from this study will be rapidly applied by physicians and public health decision makers. The results of these studies will be used as a guideline to administer zinc supplements in COVID-19 patients in order to reduce disease severity and mortality. Moreover, the experiments will clarify whether zinc supplementation as a prophylaxis strategy is useful to protect the population at risk of zinc deficiency, more than 20% worldwide. Finally, considering the new knowledge that this project will generate about the role of zinc in immune responses and viral expansion, the investigators expect that our results will help researchers and physicians to design novel strategies to boost specific immune cell subpopulations against SARS-CoV2 infection. Thus, this knowledge could be used long-term for designing medicines against SARS-CoV-2 and other viral infections.

DETAILED DESCRIPTION:
Background: The essential micronutrient zinc balances immune responses to infections and additionally directly inhibits some viruses. The investigators have recently shown a robust correlation between serum zinc levels (SZL)and COVID-19 outcome in patients and a direct effect of zinc levels on SARS-CoV-2 expansion in cell culture.These results suggest that SZL might represent an important risk factor for COVID-19 severity whose adjustment would constitute an early and cost-effective therapeutic intervention.

Objectives: To explore the therapeutic benefit of zinc supplementation for COVID-19 patients and to determine the cellular and molecular basis of the effect of zinc levels on SARS-CoV-2 infections.

Methodology: A randomized clinical trial supplementing COVID-19 patients with zinc will be carried out and viral loads, inflammatory and novel zinc-related clinical markers and SARS-CoV-2-specific T- and B-cell Responses monitored. Humanized-ACE2-mice models will be used to address causal-effect associations between zinc levels and SARS-CoV-2 infection. Infections of human Calu-3 cells will be used to decipher the direct antiviral action of zinc on SARS-CoV-2 life cycle. Expected results: The investigators will generate a clear insight into zinc functioning in COVID-19 patients that might provide a therapeutic guideline immediately applicable to reduce the severity of SARS-CoV-2 pathogenicity and possibly other virus infections.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection requiring hospital admission.

Exclusion Criteria:

* Previous immunization against SARS-CoV-2
* <18 years
* pregnancy/breastfeeding
* oral intolerance
* life expectancy <72h on admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Risk of progression | day 14
  progression to severe forms of SARS-Cov-2 disease, assessed by a combined outcome that includes mortality and/or need for ICU admission

SECONDARY OUTCOMES:
Time to clinical stability | day 14
  time until clinical stability (defined as basal saturation >94%, HR <100l/min, SBP>90mm Hg and afebrile)
hospital length of stay | day 14 and day 28
  days of hospital stay
Adverse Effects | Day 14 and Day 28
  Adverse Effects

CONTACTS AND LOCATIONS:
Overall Officials: Robert Güerri-Fernández, M.D. Ph.D., Principal Investigator — PsMar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will shared on demand and under reasonable basis

REFERENCES:
- [Background] Vogel-Gonzalez M, Tallo-Parra M, Herrera-Fernandez V, Perez-Vilaro G, Chillon M, Nogues X, Gomez-Zorrilla S, Lopez-Montesinos I, Arnau-Barres I, Sorli-Redo ML, Horcajada JP, Garcia-Giralt N, Pascual J, Diez J, Vicente R, Guerri-Fernandez R. Low Zinc Levels at Admission Associates with Poor Clinical Outcomes in SARS-CoV-2 Infection. Nutrients. 2021 Feb 9;13(2):562. doi: 10.3390/nu13020562. PMID 33572045
- [Derived] Gomez-Zorrilla S, Sendra E, Du J, Espona M, Fierro-Villegas A, Siverio A, Rodriguez-Alarcon A, Castaneda S, Lopez Montesinos I, Plata C, Arrieta-Aldea I, Soldado-Folgado J, Garcia-Giralt N, Vicente R, Guerri-Fernandez R. Zinc adjuvant treatment in SARS-CoV-2: A randomized clinical trial. J Trace Elem Med Biol. 2025 Dec;92:127778. doi: 10.1016/j.jtemb.2025.127778. Epub 2025 Oct 10. PMID 41076985

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT05778383/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT05778383/ICF_001.pdf